CLINICAL TRIAL: NCT02497599
Title: A Phase 1 Study to Evaluate the Safety and Feasibility of Intraoperative Detection of Clear Cell Renal Cell Carcinoma Using Indium-111-DOTA-girentuximab-IRDye800CW
Brief Title: Intraoperative Dual-modality Imaging in Renal Cell Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13071988
Record Dates: First submitted 2015-06-02; First posted 2015-07-14 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-03

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intraoperative dual-modality imaging (Experimental): Patients receive a single intravenous dose of Indium-111-DOTA-Girentuximab-IRDye800CW. At day 4 or 5 after antibody injection a whole body planar scan and SPECT/CT scan will be acquired. At day 7 standard of care (partial) nephrectomy will be performed. This will be extended with the use of dual-modality imaging.
  Interventions: Drug: Indium-111-DOTA-Girentuximab-IRDye800CW; Radiation: SPECT/CT; Procedure: Intraoperative dual-modality imaging

INTERVENTIONS:
Drug: Indium-111-DOTA-Girentuximab-IRDye800CW — Indium-111-DOTA-Girentuximab-IRDye800CW tracer injection will be administered 7 days before (partial) nephrectomy
  Other Names: Dual-labeled girentuximab
Radiation: SPECT/CT — 4 or 5 days after tracer injection a SPECT/CT of the abdomen will be acquired.
Procedure: Intraoperative dual-modality imaging — 7 days after dual-labeled girentuximab injection standard of care surgery will be performed extended with the use of dual-modality imaging.
  Other Names: Fluorescence and radioguided surgery

SUMMARY:
Intraoperative tumor localization and resection can be enhanced using intraoperative fluorescence imaging and radiodetection. Girentuximab specifically recognizes carbonic anhydrase IX expressed on > 95% of renal cell carcinoma (RCC). Therefore Indium-111-DOTA-girentuximab-IRDye800CW is a perfect dual-labeled antibody for dual-modality image-guided surgery in RCC.

The aim of this study is to assess the feasibility and safety of intraoperative dual-modality imaging with Indium-111-DOTA-girentuximab-IRDye800CW in renal cell carcinoma patients.

DETAILED DESCRIPTION:
In oncologic surgery complete tumor resection is important for treatment outcome and patient survival. Intraoperative tumor localization and resection can be enhanced using intraoperative imaging techniques (e.g. targeted radioguided or fluorescence guided surgery). A powerful synergy can be achieved by combining radiotracers (e.g. Indium-111) and optical tracers (e.g. IRDye 800CW) conjugated to an antibody against a tumor-associated antigen. Girentuximab specifically recognizes carbonic anhydrase IX expressed on > 95% of renal cell carcinoma (RCC). Therefore Indium-111-DOTA-girentuximab-IRDye800CW is a perfect dual-labeled antibody for dual-modality image-guided surgery in RCC. The concept has been shown in preclinical studies with mice and the investigators will translate this to the clinic.

Eligible patients with renal cell carcinoma scheduled for (partial) nephrectomy will receive dual-labeled girentuximab 7 days before surgery. At day 4 or 5 a SPECT/CT of the abdomen will be obtained. Surgery at day 7 will be extended with the use of a near-infrared fluorescence camera and a gamma probe.

The aim of this study is to assess the feasibility and safety of intraoperative dual-modality imaging with Indium-111-DOTA-girentuximab-IRDye800CW in renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of clear cell renal cell carcinoma planned for surgery, (partial) nephrectomy
* Performance status: Karnofsky 70 %
* Being fit for surgery
* Minimum age 18 years
* Signed informed consent

Exclusion Criteria:

* A known subtype other than clear cell RCC
* Any medical condition present that in the opinion of the investigator will affect patients' clinical status.
* Administration of a radioisotope within 10 physical half lives prior to study enrollment
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Fluorescent signal at time of surgery | During surgery
  Can the tumor be identified by the fluorescent signal? Yes/No. Can the tumor be distinguished from normal tissue? Yes/No

SECONDARY OUTCOMES:
Safety of dual-labeled antibody injection as assessed by the number of participants with grade 3 or 4 Adverse Events according to CTCAE v4.0 | 4 weeks
  The number of participants with grade 3 or 4 Adverse Events according to CTCAE v4.0 will be scored.
Blood levels of the dual-labeled antibody | 60, 120 and 180 minutes after injection and 4 and 7 days after injection
  Blood samples will be measured for radioactivity in a gamma counter at different timepoints after injection. This will be expressed as percentage injected dose per gram (%ID/g).
Optimal dose of the dual-labeled antibody preparation | 4 weeks
  Tumor to background ratio will be evaluated for each dose.

CONTACTS AND LOCATIONS:
Overall Officials: Peter FA Mulders, M.D. PhD, Principal Investigator — Radboud University Medical Center; Wim JG Oyen, M.D. PhD, Study Director — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No